CLINICAL TRIAL: NCT05582603
Title: Detailed Study on the Safety, Dosage and Feasibility of an Intervention Based on a Computerized Cognitive Training (CCT) for Individuals With Post-acute Sequelae of COVID-19 (PASC): A Phase I/II Trial
Brief Title: Safety and Dosage of a Computerized Cognitive Training Program for Cognitive Dysfunction After COVID-19
Acronym: CCTLongCOVID
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Antonio de Nebrija (Other)
Responsible Party: Principal Investigator, Jon Andoni Duñabeitia, Director of Research Center, Universidad Antonio de Nebrija
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNNE-2021-010
Record Dates: First submitted 2022-10-13; First posted 2022-10-17 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Post-Acute COVID-19; Post Acute COVID-19 Syndrome; Cognitive Dysfunction; Cognitive Impairment
Keywords: post-acute sequelae of COVID-19; PASC; cognitive dysfunction; computerized cognitive training; brain training
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Phase I: An open-label prospective Phase I dose-escalation study following a standard 3+3 rule-based up-and-down design without dose de-escalation will be followed.
  Phase II: An open-label prospective clinical trial to validate the minimum dosage and appropriate safety using the training time obtained in Phase I for the CCT along a 15-day training period with a 24-hour rest between sessions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Computerized Cognitive Training (Experimental): Individuals enrolled in Phase I and II will complete a Computerized Cognitive Training (CCT) based on an intervention with 15 different cognitive tasks in the form of games aimed at enhancing memory, attention, reasoning, perception and coordination skills. The CCT will be implemented in an app designed by CogniFit (CogniFit Inc., San Francisco, USA) to be used in tablets or mobile phones.
  Interventions: Behavioral: CCT Long COVID

INTERVENTIONS:
Behavioral: CCT Long COVID — A 15-day training protocol in which every 48 hours participants' complete a series of different cognitive tasks in the form of games selected among a pool of 12 games from CogniFit (CogniFit Inc., San Francisco, USA) whose difficulty level is tailored to each individual by the a patented Individualized Training System™ (ITS) software that automatically chooses the activities and difficulty levels for each person in every session.
  Other Names: CogniFit CCT Long COVID

SUMMARY:
The goal of this Phase I/II clinical trial is to assess the safety and maximum tolerated training time of a self-administered computerized cognitive training (CCT) in individuals with cognitive dysfunction as a consequence of COVID-19 infection.

DETAILED DESCRIPTION:
A Phase I/II protocol is designed to determine the safety of a Computerized Cognitive Training (CCT) aimed at ameliorating the cognitive dysfunction often observed in persons with post-acute sequelae of COVID-19 (PASC). The Phase I/II trial also aims at establishing the maximum tolerated training time per session of the CCT and to explore the feasibility of such intervention. In Phase I, through a 3+3 design, a dose-escalation trial will be set. Participants will be tested across subsequent training blocks of 15 minutes each, reporting on the experienced fatigue or adverse effects after every block. The safe training dose will be set to a block before extreme fatigue or a notable adverse effect has been reported by two or more participants. Once a safety training time has been established, a group of participants will engage in a 15-day training effectiveness assessment. After an initial thorough pre-test assessment, the intervention protocol will start. An evaluation day and a training day will be interspersed so that participants will complete a total of 8 training sessions (days 1, 3, 5, 7, 9, 11, 13 and 15). After the final day of intervention, a post-test assessment session will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 25 and 55 years old.
* History of infection with COVID-19 at least 3 months prior to expression of interest with a valid diagnostic or antibody test.
* Presence of self-perceived cognitive dysfunction associated with post-acute sequelae of COVID-19 (concentration problems or brain fog).

Exclusion Criteria:

* Suicidal traits.
* Poor digital skills.
* Not having access to a mobile phone or tablet with Internet connection during the time of the intervention (only for Phase II).
* Not having 60 spare minutes per day to complete the intervention (only for Phase II).

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-10-18 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Fatigue Level Questionnaire | In Phase I, after each iteration of a 15-minute training.
  Fatigue questionnaire adapted from the Brief Fatigue Inventory (Mendoza et al., 1999)
Fatigue Level Questionnaire | In Phase II, on even days (rest days of the intervention protocol).
  Fatigue questionnaire adapted from the Brief Fatigue Inventory (Mendoza et al., 1999)
Safety Level Questionnaire | In Phase I, after each iteration of a 15-minute training.
  Safety questionnaire aimed at exploring the existence of side effects and/or adverse events.
Safety Level Questionnaire | In Phase II, on even days (rest days of the intervention protocol).
  Safety questionnaire aimed at exploring the existence of side effects and/or adverse events.
Classification of side effect or adverse events | In Phase I, after each iteration of a 15-minute training, only in case side effects or adverse events have been reported in the Safety Questionnaire.
  Interview adapted from the Patient-Reported Adverse Drug Event Questionnaire (de Vries et al., 2013).
Classification of side effect or adverse events | In Phase II, on even days (rest days of the intervention protocol), only in case side effects or adverse events have been reported in the Safety Questionnaire.
  Interview adapted from the Patient-Reported Adverse Drug Event Questionnaire (de Vries et al., 2013).

SECONDARY OUTCOMES:
Computerized Cognitive Assessment | In Phase II, at pre-test (the day before the intervention protocol starts) and at post-test (the day after the intervention protocol finishes).
  Complete cognitive evaluation based on Cognitive Assessment Battery (CogniFit Inc., San Francisco, USA).
Quality of Life Assessment | In Phase II, at pre-test (the day before the intervention protocol starts) and at post-test (the day after the intervention protocol finishes).
  Short version of the self-perceived global physical and mental health scale from the Patient-Reported Outcomes Measurement Information System (PROMIS v.1.2).
Paper-and-pencil Cognitive Assessment | In Phase II, at pre-test (the day before the intervention protocol starts) and at post-test (the day after the intervention protocol finishes).
  The Montreal Cognitive Assessment (MoCA).

CONTACTS AND LOCATIONS:
Overall Officials: Jon Andoni Duñabeitia, PhD, Principal Investigator — Universidad Nebrija
Locations (1):
- Universidad Nebrija, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No